CLINICAL TRIAL: NCT05084092
Title: IORT After Surgical Resection of Brain Metastases: Feasibility and Efficacy Phase II Trial
Brief Title: IORT After Surgical Resection of Brain Metastases
Acronym: IORT_BRAINM1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IORT_BRAIN_MET_2019
Record Dates: First submitted 2021-04-08; First posted 2021-10-19 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Brain Neoplasms
Keywords: Brain metastases; neurosurgery; intraoperative radiotherapy; local therapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Intraoperative Radiation Therapy (IORT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Radiotherapy (IORT) (Experimental): Intraoperative Radiotherapy (IORT) administered during surgery
  Interventions: Radiation: Intraoperative Radiotherapy (IORT); Procedure: Brain surgery

INTERVENTIONS:
Radiation: Intraoperative Radiotherapy (IORT) — If biopsy is positive, local treatment with IORT will be performed. After IORT (15,40 Gray at 2 mm dept), the applicator will be removed and surgery will be continued in a standard fashion.
Procedure: Brain surgery — Surgery should be performed according to the local standard of care, preferentially as image-(neuronavigation) guided surgery. To establish the diagnosis of a metastasis and to exclude primary CNS tumors, lymphomas, SCLCs or germinomas it will be performed a peroperative biopsy

SUMMARY:
To evaluate the feasibility and efficacy of the Intraoperative Radiation Therapy (IORT) after the resection of a brain metastases to reduce the incidence of local relapse

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, Karnofsky Performance Index ≥ 70.
* Newly diagnosed cerebral or cerebellar lesion (contrast enhancing on a T1- weighted MRI scan) amenable to total resection with no dural attachment.
* Frozen section confirming a metastasis of an extracranial (i.e. non-CNS) tumor.
* Adequate distance to optic nerve(s), chiasm and brainstem (organs at risk for radiotherapy).
* Adequate birth control.
* Informed consent.

Exclusion Criteria:

* Leptomeningeal spread and dural attachment (assessed pre- and intraoperative).
* Frozen section reveals primary CNS tumor, lymphoma, SCLC or germinoma.
* Psychiatric or social condition potentially interfering with compliance.
* Contraindication against anesthesia, surgery, MRI and/or contrast agents.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Median local progression free survival (PFS) | 12 months
  Time span (in months) between surgery and recurrence within a 0,5 cm margin around the resection cavity, evaluated through Response Assessment in Neuro-Oncology (RANO) criteria for brain metastasis obtained from serial Magnetic resonance imaging (MRI) scans.

SECONDARY OUTCOMES:
Median regional PFS (rPFS) | 12 months
  The time (in months) from surgery to any progression outside of the 0,5 cm margin around the resection cavity, evaluated through Response Assessment in Neuro-Oncology (RANO) criteria for brain metastasis obtained from serial Magnetic resonance imaging (MRI) scans.
Global PFS (gPFS) | 12 months
  Time (in months) from surgery to any intra- and extracranial tumor progression evaluated through Response Assessment in Neuro-Oncology (RANO) criteria for brain metastasis obtained from serial Magnetic resonance imaging (MRI) scans.
Median time to the initiation of systemic therapies | 12 months
  Time (in days) from surgery to the day of initiation of any systemic anti-tumor therapy (e.g., chemotherapy)
Median overall survival (OS) | 12 months
  Time (in months) from surgery of brain metastases to death by any cause
Change in neurocognitive performance (compared to baseline): Minimental | 6, and 12 months
  Assessed by minimal mental scale examination
Change in neurocognitive performance (compared to baseline): Trail making | 6, and 12 months
  Assessed by trail making test
Change in neurocognitive performance (compared to baseline): Repetition | 6, and 12 months
  Assessed by number repetition test (forward and backward)
Change in neurocognitive performance (compared to baseline): Oral | 6, and 12 months
  Assessed by controlled oral word association test
Change in neurocognitive performance (compared to baseline): Semantic | 6, and 12 months
  Assessed by semantic word association
Quality of life (QoL) | 6, and 12 months
  Assessed by European Organization for Research and Treatment (EORTC)- Quality of Life Questionnaires (QLQ C30/BN20)
Radiation-related (acute / early delayed / late) neurotoxicity | 12 months
  Assessed by regular neurological examinations combined by serial MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Macià, MD, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Catalan Institute of Oncology, L'Hospitalet de Llobregat, Barcelona, Spain